CLINICAL TRIAL: NCT02169921
Title: Determination of Safety and Effectiveness of the TurboHawk and the SpiderFX for the Treatment of Peripheral Arterial Disease in the Superficial Femoral and/or the Popliteal Arteries in Japan
Brief Title: TurboHawk™ Japan Trial in Patients With PAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVJ-12-02-01
Record Dates: First submitted 2014-06-08; First posted 2014-06-23 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TurboHawk (Experimental): This study is designed as a single arm study. For angioplasty, the Atherectomy Catheter, TurboHawk is used in this arm. Spider FX, the Distal Embolus Protection Device, can concomitantly be used with TurboHawk
  Interventions: Device: Atherectomy Catheter

INTERVENTIONS:
Device: Atherectomy Catheter — Atherectomy Catheter, TurboHawk, is used for Angioplasty. Spider FX can concomitantly be used with TurboHawk.
  TurboHawkTM LS-C, TurboHawk LX-C, TurboHawk SS-CL and TurboHawk SX-C are participated in this arm.

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the TurboHawk for the treatment of peripheral arterial disease (PAD) in the superficial femoral and/or the popliteal arteries with the Japanese population.

ELIGIBILITY:
Inclusion Criteria:

* Provides written informed consent
* Willing to comply with follow-up evaluations at specified times
* Has a Rutherford Clinical Category Score of 2-4
* Disease located within the femoropopliteal artery
* Has evidence of ≥ 50% stenosis or occlusion in the superficial femoral and/or popliteal, confirmed by angiography
* Each discrete target lesion's length is ≥4cm and ≤ 15 cm
* Reference vessel diameter is ≥ 3.5 mm and ≤ 7.0 mm

Exclusion Criteria:

* Previously implanted stent(s) or stent graft(s) in target leg
* Life expectancy less than 12 months
* Has any planned surgical or endovascular intervention of target vessel 30 days before or after index procedure
* Has in-stent restenosis of the target lesion
* Has an aneurysmal target vessel
* Has perforation, dissection or other injury of the access or target vessel requiring additional stenting or surgical intervention prior to enrollment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-06; Primary Completion 2015-09 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Primary Patency Rate | 180 Days

SECONDARY OUTCOMES:
Technical procedural success | 30 Days
Preservation of the number of run-off vessels determined by angiography | intra operative
Event free survival | 30 Days , 180 Days and One Year
Amputation Rate | 30 Days , 180 Days and One Year
Improvement in Rutherford Clinical Category | 30 Days , 180 Days and One Year
Improvement in Ankle-Brachial Index | 30 Days , 180 Days and One Year
Clinically driven target lesion revascularisation | 30 Days , 180 Days and One Year
Clinically driven target vessel revascularisation | 30 Days , 180 Days and One Year

CONTACTS AND LOCATIONS:
Overall Officials: Takao Ohki, MD, Principal Investigator — Jikei University School of Medicine; Hiroshi Ando, MD, Principal Investigator — Kasukabe Chuo General Hospital
Locations (2):
- Japan (2):
  - Kasukabe Chuo General Hospital, Kasukabe, Saitama
  - Jikei University School of Medicine, Minato-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Undecided